CLINICAL TRIAL: NCT01558869
Title: An Open-label, Single-centre, Single-arm Phase II Study of Capecitabine Combined With Oxaliplatin and Irinotecan (Xeloxiri) as First-line Treatment in Patients With Advanced Unresectable Pancreatic Adenocarcinoma
Brief Title: Xeloxiri as First-line Treatment in Patients With Advanced Unresectable Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. YAU Chung Cheung Thomas, Clinical Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MONC-HBP24
Record Dates: First submitted 2012-03-18; First posted 2012-03-20 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Pancreatic Adenocarcinoma
MeSH Terms: interventions — Capecitabine; Oxaliplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Drug: Irinotecan

INTERVENTIONS:
Drug: Capecitabine — 1200 mg/m2 BD orally for 1 week of a 2-week cycle (i.e. 1 week on, 1 week off)
  Other Names: Xeloda
Drug: Oxaliplatin — 70 mg/m2 IV on day 1 of a 2-week cycle
Drug: Irinotecan — 130 mg/m2 IV on day 1 of a 2-week cycle

SUMMARY:
This is an open-label, single centre, single-arm phase II study which aims to assess the efficacy and tolerability of triplet combination of capecitabine, oxaliplatin and irinotecan (Xeloxiri regimen) in treating patients with advanced unresectable pancreatic carcinoma. Clinical data from patients diagnosed with pancreatic adenocarcinoma will be collected and analyzed in this study. The patients' data will be collected and maintained in the Division of Medical Oncology of the University Department of Medicine, Queen Mary Hospital, Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age, male or female.
* Histopathologically or cytologically confirmed adenocarcinoma of the pancreas.
* ECOG performance status 0 to 2.
* Adequate bone marrow reserve.
* Absolute neutrophil count > 1x10^9/L.
* Total bilirubin <3 times the upper limit of the normal range.
* Life expectancy ≥ 12 weeks.
* Signed written informed consent form.

Exclusion Criteria:

* Prior malignant disease other than pancreatic cancer.
* Patients suitable for surgical or locoregional therapies.
* Patients who have prior anticancer therapy for pancreatic cancer.
* Patients unable to swallow oral medications.
* Any evidence of brain metastasis (unless the patient is >6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry).
* Active clinically serious infections (> grade 2 NCI / CTC Adverse Event version 3.0).
* History of allergy to platinum compounds.
* Patients who have chronic inflammatory bowel disease and/or bowel obstruction.
* Patients who have severe bone marrow failure.
* Patients undergoing renal dialysis.
* History of HIV infection.
* Seizure disorder requiring medication (such as steroids or anti-epileptics).
* Women who are pregnant or breast-feeding, or women of child-bearing potential who are unable or unwilling to practice a highly effective means of contraception.
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in extent of disease | Change from baseline in size approximately every 4 cycles
  Objective response rate

SECONDARY OUTCOMES:
CA19.9 reduction | Change from baseline every 2 cycles
Progression-free survival | From date of start until the date of first documented progression or death from disease-related causes or last follow-up, whichever came first, assessed up to 18 months
Overall survival | From date of start until the date of death from any cause or last follow-up, whichever came first, assessed up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Yau, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, The University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347